CLINICAL TRIAL: NCT02984488
Title: Post-Obturation Pain Following One-visit Versus Two-visit Root Canal Treatment of Necrotic Anterior and Premolar Teeth Using Protaper Next
Brief Title: Pain Following One-visit Versus Two-visit Root Canal of Necrotic Teeth Using Protaper Next
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hebatallah Mostafa Mahmoud Ahmed Nada, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: single_two visits
Record Dates: First submitted 2016-11-14; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-11

CONDITIONS: Tooth, Nonvital
Keywords: necrotic teeth; single visit; multiple visits; protaper next
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- single visit endodontic treatment. (Experimental): •single visit endodontic Treatment of necrotic teeth using Protaper next.
  Interventions: Procedure: single visits
- Two visits endodontic treatment (Active Comparator): •Two visits endodontic Treatment of necrotic teeth using Protaper next.
  Interventions: Procedure: two visits

INTERVENTIONS:
Procedure: single visits — Endodontic treatment is done and completed in a single visit using protaper next rotary system.
  Arms: single visit endodontic treatment.
Procedure: two visits — Endodontic treatment is done and completed in two visits using protaper next rotary system.
  Arms: Two visits endodontic treatment

SUMMARY:
To evaluate the incidence and severity of postoperative pain after root canal therapy of necrotic teeth in one appointment versus two appointments using Protaper next instrument.

DETAILED DESCRIPTION:
The key to endodontic success was described as the debridement and neutralization of any tissue, bacteria, or inflammatory products within the root canal system.

Endodontic treatment used to take multiple visits to complete, with one of the main reasons for this being that it required a considerable amount of time to complete the treatment.

The single-visit treatment was bought back in the 1950s by Ferranti, who advocated the use of diathermy for pulpal disinfection and hydrogen peroxide for irrigation.

The use of contemporary endodontic techniques and equipment, such as use of rubber dam, magnifying devices, electronic apex locators, engine-driven rotary nickel titanium files, and so forth, not only increases the success rate of endodontic treatment but also, shortens the time needed for the treatment. Endodontic treatment may therefore be completed in a single visit.

It is generally agreed upon that the prepared canals can never be sterile before obturation, no matter how potent the antibacterial irrigants or intracanal medications are. There are currently two measures to reduce bacterial persistence and reinfection in the canals. We can either dress the canals with antibacterial agents in multiple visits or immediately obturate the canals, to reduce the space for bacterial colonization, in a single-visit approach. Calcium hydroxide is the most commonly used intracanal medicament, however its efficacy towards Enterococcus faecalis is questionable.

ELIGIBILITY:
Inclusion criteria:

* Medically free patients.
* Patient's age above 18 years old.
* Teeth diagnosed clinically with necrosis.
* Positive patient's acceptance for participation in the study.
* Sex includes both male and female.
* Patients who can understand visual analogue scale.
* Patients able to sign informed consent.

Exclusion criteria:

* Pregnancy or lactation.
* Medically compromised patients.
* Patient with multiple teeth that required treatment in the same quadrant to eliminate the possibility of pain referral.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Change of post operative pain. | After 6-12-24-48 hours from the obturation step of the endodontic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Saeed M Abd El aziz, professor, Study Chair — Department of endodontics - Faculty of Oral and Dental medicine - CU; hebatallah M nada, student, Principal Investigator — Department of endodontics - Faculty of Oral and Dental medicine - CU

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rao KN, Kandaswamy R, Umashetty G, Rathore VP, Hotkar C, Patil BS. Post-Obturation pain following one-visit and two-visit root canal treatment in necrotic anterior teeth. J Int Oral Health. 2014 Apr;6(2):28-32. Epub 2014 Apr 26. PMID 24876699
- [Background] DiRenzo A, Gresla T, Johnson BR, Rogers M, Tucker D, BeGole EA. Postoperative pain after 1- and 2-visit root canal therapy. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2002 May;93(5):605-10. doi: 10.1067/moe.2002.121900. PMID 12075212